CLINICAL TRIAL: NCT04538209
Title: Assessment of Portal Circulation Before and After Variceal Eradication in Patients With Liver Cirrhosis.
Brief Title: Effect of Variceal Eradication on Portal Circulation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Yousef Mohammed, Assistant Lecturer of Tropical Medicine and Gastroenterology, Assiut University
Other Study IDs: portal circulation assessment
Record Dates: First submitted 2020-08-30; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Portosystemic Collateral Veins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- canditates for variceal eradication: patients with documented liver cirrhosis (Based on clinical, laboratory and ultrasonographic findings) undergoing either primary or secondary prophylaxis variceal eradication at endoscopy unit of El-Rajhi hospital, Assuit University
  Interventions: Radiation: Abdominal computed tomography with angiography.

INTERVENTIONS:
Radiation: Abdominal computed tomography with angiography. — technique of combing a Computed Tomography scan with the injection of dye to create pictures of the portal circulation and portosystemic collaterals veins.

SUMMARY:
Study the effect of variceal eradication on portal circulation, liver stiffness and Child-Pugh and MELD scores in patients with liver cirrhosis.

DETAILED DESCRIPTION:
Portosystemic collateral circulation is a consequence of portal hypertension, which occurs in chronic liver disease and is responsible for numerous complications.

Gastric and oesophageal varices are two of common portosystemic collaterals, patients usually presented with hematemesis, melena, or both, ultimately 20% is the mortality during the first attack.

Although both band ligation and sclerotherapy are effective modalities of treatment in controlling acute variceal bleeding, in preventing future variceal bleeding as well as in eradicating varices with very few complications , their effects on portal circulation have raised concerns among hepatologist.

Information about collateral pathways is especially relevant when interventional procedures or surgery is indicated because inadvertent distribution of these vessels can cause significant bleeding.

Few studies pointed on development of new portosystemic collaterals post variceal eradication depending on abdominal computed tomography (CT ) compared to pre-variceal eradication as showed paraoesophageal varices, retro-gastric varices not visualized with endoscopy ,or large deep gastric collaterals that may increase risk for rebleeding.

Also, liver stiffness measurement and indirect markers of portal hypertension have been correlated with the severity of portal hypertension and have been used to predict the presence of varices, and there is rising question what about effect of variceal eradication on liver stiffness.

The Child-Pugh and MELD scores were significantly higher for patients with gastric variceal bleeding , and the question here is variceal eradication can improve Child-Pugh and MELD scores or there is no effect.

ELIGIBILITY:
Inclusion Criteria:

* • Age between 18 and 70 years old.

  * Patient with documented liver cirrhosis undergoing either primary or secondary prophylactic variceal eradication.
  * Liver cirrhosis with Child-Pugh score A and B.

Exclusion Criteria:

* • Age less than 18 years.

  * Have contraindications to computed abdominal CT-angiography (e.g. allergy to all suitable contrast agents, renal failure).
  * Patients with history of recent significant bleeding varices.
  * Previous history of variceal ligation, sclerotherapy, and TIPS operation.
  * Patients with isolated gastric varices.
  * Patients with HCC or other malignancies.
  * End-stage liver disease (Child score more than 9).
  * Patients with malignant portal vein thrombosis.
  * Patients with non-cirrhotic portal hypertension.
  * Patients refuse to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with documented liver cirrhosis (Based on clinical, laboratory and ultrasonographic findings) undergoing either primary or secondary prophylaxis variceal eradication at endoscopy unit of El-Rajhi hospital, Assuit University.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Study the effect of variceal eradication on portal circulation, liver stiffness and Child-Pugh and MELD scores in patients with liver cirrhosis. | 4 years
  Study the effect of variceal eradication on portal circulation and development of new portosystemic collaterals had not be found before variceal eradication in patients with liver cirrhosis

SECONDARY OUTCOMES:
Study the effect of variceal eradication on liver stiffness and Child-Pugh and MELD scores in patient with liver cirrhosis | 4 years
  study how can variceal eradication affect liver elasticity, liver function so can calculate Child-Pugh and MELD scores which can life expectancy of patients with liver cirrhosis

CONTACTS AND LOCATIONS:
Overall Officials: Esraa Swifee, Principal Investigator — Assiut University

REFERENCES:
- [Background] Abdel-Aty M, Fouad M, Sallam MM, Elgohary EA, Ismael A, Nawara A, Hawary B, Tag-Adeen M, Khaled S. Incidence of HCV induced-Esophageal varices in Egypt: Valuable knowledge using data mining analysis. Medicine (Baltimore). 2017 Jan;96(4):e5647. doi: 10.1097/MD.0000000000005647. PMID 28121921
- [Background] Garcia-Tsao G, Abraldes JG, Berzigotti A, Bosch J. Portal hypertensive bleeding in cirrhosis: Risk stratification, diagnosis, and management: 2016 practice guidance by the American Association for the study of liver diseases. Hepatology. 2017 Jan;65(1):310-335. doi: 10.1002/hep.28906. Epub 2016 Dec 1. No abstract available. PMID 27786365
- [Background] Augustin S, Millan L, Gonzalez A, Martell M, Gelabert A, Segarra A, Serres X, Esteban R, Genesca J. Detection of early portal hypertension with routine data and liver stiffness in patients with asymptomatic liver disease: a prospective study. J Hepatol. 2014 Mar;60(3):561-9. doi: 10.1016/j.jhep.2013.10.027. Epub 2013 Nov 6. PMID 24211744
- [Background] Lahbabi M, Mellouki I, Aqodad N, Elabkari M, Elyousfi M, Ibrahimi SA, Benajah DA. Esophageal variceal ligation in the secondary prevention of variceal bleeding: Result of long term follow-up. Pan Afr Med J. 2013 May 3;15:3. doi: 10.11604/pamj.2013.15.3.2098. Print 2013. PMID 23847700